CLINICAL TRIAL: NCT06703398
Title: A Multicenter, Randomized, Controlled,Open Label, Phase II Trial of Autologous Tumor Infiltrating Lymphocytes (GC101 TIL) in Subjects With Advanced Melanoma
Brief Title: A Study of GC101 TIL in Advanced Melanoma
Acronym: MIZAR-003
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC101 TIL-MM-II
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Randomized-controlled trial; Tumor Infiltrating Lymphocytes; Chemotherapy
MeSH Terms: conditions — Melanoma | interventions — Dacarbazine; Temozolomide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC101 TIL group (Experimental): A tumor sample is resected from each participant and cultured ex vivo to expand the population of autologous tumor infiltrating lymphocytes injection (GC101 TIL). After lymphodepletion, patients are infused GC101 TIL followed sintilimab.
  Interventions: Biological: GC101 TIL
- Investigator's choice of chemotherapy (Active Comparator): monotherapy or combination of dacarbazine, temozolomide, paclitaxel,carboplatin or cisplatin, and the chemotherapy's dosage could refer to the drug label or the relevant treatment guideline, the final decision is up to investigator.
  Interventions: Drug: dacarbazine, temozolomide, paclitaxel ,platinum or cisplatin

INTERVENTIONS:
Biological: GC101 TIL — Patients with advanced melanoma (excluding uveal melanoma) who have failed to PD-1 antibodies (if BRAF mutation is present, BRAF and MEK inhibitors have failed; if NRAS mutation is present, tunlametinib have failed) and are ineligible for resection
  Arms: GC101 TIL group
Drug: dacarbazine, temozolomide, paclitaxel ,platinum or cisplatin — monotherapy or combination of dacarbazine, temozolomide, paclitaxel, platinum or cisplatun, and the chemotherapy's dosage could refer to the drug label or the relevant treatment guideline, the final decision is up to investigator
  Arms: Investigator's choice of chemotherapy

SUMMARY:
98 participants will be randomly assigned 1:1 to the experimental group and the control group for the Phase II clinical trial，this trail is expected to be finished in 24 months

DETAILED DESCRIPTION:
This study is to investigate the efficacy and safety of autologous tumor infiltrating lymphocyte (GC101 TIL) therapy versus investigator's choice of chemotherapy in patients with advanced melanoma. Autologous TILs are expanded from tumor resections or biopsies and infused i.v. into the patient after NMA lymphodepletion treatment with cyclophosphamide and hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF) and able to comply with the visits and related procedures specified in the protocol;
* Aged ≥18 years and ≤75 years, regardless of gender;
* Patients with unresectable advanced, recurrent or metastatic melanoma (excluding uveal melanoma) ;
* Patients who have failed or resisted to PD-1 antibodies；
* Patients must have failed or resisted to at least two frontlines systemic tehrapy(if knowed with BRAF V600 mutate, then need to failed to BRAF/MEK inhibitor; if knowed with NRAS mutate, then need to failed to Tunlametinib) ；
* TILs can be isolated from a surgically resectable tumor region: the tissue volume must be >150mm3, and the lesion has not received local treatment (such as radiotherapy, radiofrequency ablation, oncolytic virus, etc.) or progressed after local treatment;There are still at least 1 measurable lesion (according to RECIST1.1 criteria ) even after TIL sampling and resection of surgically resectable tissue;
* ECOG performance status 0-1;
* Expected survival time >3 months;
* With sufficient hematology and end-organ function;
* Good compliance and able to adhere to the study visit plan and other agreement requirements.

Exclusion Criteria:

* Patients receive any drug under study within 28 days prior to screening;
* Combination of 2 or more malignant tumors, except: Eradicated malignant tumors that have been inactive for ≥5 years prior to study entry and are at minimal risk of recurrence; adequately treated non-melanoma skin cancer or malignant nevus of freckle-like nevus without evidence of disease recurrence; adequately treated carcinoma in situ without evidence of disease recurrence;
* Has received live attenuated vaccination after signing informed consent or is scheduled to receive it during the study;
* Has not recovered from a prior procedure or treatment-related adverse reaction to ≤ grade 1 nci ctcae 5.0 (except for toxicities such as alopecia, hypothyroidism etc., which in the judgment of the investigator pose no safety risk);
* Known history of allergy to streptomycin, ciprofloxacin, or micafungin or allergy to any component of the infused product formulation;
* Uncontrolled co-morbidities including, but not limited to, uncontrolled arterial hypertension (systolic blood pressure ≥160 mmhg and/or diastolic blood pressure ≥100 mmhg) even with standardized treatment or any unstable cardiovascular disease including transient ischemic attack, cerebrovascular accident, myocardial infarction, unstable angina pectoris within 6 months prior to enrollment; new york heart association ( nyha class iii or iv congestive heart failure with an ejection fraction <50%; or severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias, degree ii-iii atrioventricular block, etc., requiring clinical intervention; ecg results showing clinically significant abnormalities or a qtcf ≥450ms (if the first test is abnormal, it may be retested at least 5 minutes apart twice and the combined result/mean value to determine eligibility) ;
* Patients with esophageal or gastric varices that require immediate intervention (e.g., taping or sclerotherapy) or are considered to be at high risk for bleeding based on the opinion of the investigator or consultation with a gastroenterologist or hepatologist, have evidence of portal hypertension (including splenomegaly detected on imaging), or have a prior history of variceal bleeding must have undergone endoscopic evaluation within 3 months prior to enrollment;
* Uncontrolled metabolic disorders, such as diabetes mellitus known to be uncontrolled, or other non-malignant organ or systemic diseases or secondary reactions to cancer, and which can lead to higher medical risk and/or uncertainty in survival evaluation;
* Hepatic encephalopathy, hepatorenal syndrome or child-pugh class b or more severe cirrhosis, liver failure;
* With other serious organic diseases or mental disorders;
* Suffering from systemic active infection requiring treatment, with positive blood culture or imaging evidence of infection, including but not limited to active tuberculosis;
* Suffering from infectious diseases such as hepatitis B, hepatitis C, syphilis, AIDS, etc;
* Individuals with active autoimmune diseases (such as eczema, vitiligo, psoriasis, alopecia or Graves' disease that do not require systemic treatment within the past two years, other autoimmune diseases that are not expected to recur, hypothyroidism that only requires thyroid hormone replacement therapy, and type 1 diabetes that only requires insulin replacement therapy can be enrolled);
* Any NCI CTCAE 5.0 immune-related adverse reaction (iRAE) grade ≥3 occurred during any previous immunotherapy(except for cases where it recovered to ≤1 after treatment or reached stability as assessed by the investigator);
* Those who had undergone organ allotransplantation, allogeneic stem cell transplantation and renal replacement therapy;
* Pulmonary fibrosis, interstitial lung disease (including past history and current condition), acute lung disease;
* Those with leptomeningeal metastasis;
* Patients with clinical symptoms of central nervous system metastases (such as cerebral edema, requiring hormone intervention, or progression of brain metastases), Patients who have previously received treatment for brain metastases, such as those who have maintained clinical stability (MRI) for at least 2 months and have stopped systemic hormone therapy (dose > 10mg/ day prednisone or other equivalent hormones) for more than 4 weeks, can be included;
* Women who are pregnant or breastfeeding;
* There is a history of TIL cell therapy, allogeneic T cell therapy, or NK cell therapy within 6 months;
* Situations that are not suitable for enrollment assesed by investigators;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Every 6 weeks for 12 months
  Progression-free survival (PFS) confirmed by the Independent Review Committee (IRC) according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival | Maximum 2 years
  Overall survival (OS) and OS rates at 6, 12, and 18 months
Progression-free survival | Every 6 weeks for 12 months
  PFS assessed by investigators according to RECIST 1.1 and PFS assessed by IRC and investigators according to iRECIST
Objective Response Rate | Maximum 360 days
  Objective Response Rate (ORR) assessed by IRC and investigators according to RECIST 1.1 and iRECIST
Disease Control Rates | Every 6 weeks for 12 months
  Disease Control Rates (DCR) assessed by IRC and investigators according to RECIST 1.1 and iRECIST
Duration of Response | Every 6 weeks for 12 months
  Duration of Response (DoR) assessed by IRC and investigators according to RECIST 1.1 and iRECIST
Adverse Events | Maximum 360 days
  Incidence of adverse events associated with GC101 TIL retransfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No